CLINICAL TRIAL: NCT03332420
Title: A Real-world Study to Evaluate the Efficacy of Huaiqihuang Granule in Children With Primary Nephrotic Syndrome
Brief Title: The Efficacy of Huaiqihuang Granule in Children With Primary Nephrotic Syndrome
Status: Completed | Type: Observational
Sponsor: Qidong Gaitianli Medicines Co., Ltd (Industry)
Collaborators: Capital Institute of Pediatrics, China (Other)
Responsible Party: Sponsor
Other Study IDs: HQH-201705
Record Dates: First submitted 2017-10-15; First posted 2017-11-06 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Nephrotic Syndrome
Keywords: Huaiqihuang granule; primary nephrotic syndrome; multisite; prospective; open-label
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Observational 1: Huaiqihuang Granule
- Observational 2: Standard treatment+Huaiqihuang Granule
- Observational 3: Standard treatment

SUMMARY:
This is a multisite, open-label, prospective and registered study designed to evaluate the efficacy and safety of Huai-Qi-Huang granule in children with primary nephrotic syndrome.

DETAILED DESCRIPTION:
This is a multisite, open-label, prospective and registered study designed to evaluate the efficacy and safety of Huai-Qi-Huang granule in children with primary nephrotic syndrome(PNS). The study will be Planned at 1500 participants, and subjects will be on study for up to one year. Data will be collected by authorized physicians for 48 weeks. all of the data included demographic characteristics, information about PNS, laboratory tests and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. In accordance with Pediatric Branch , the Chinese Medical Association in 2009: guidelines for diagnosis and treatment of common kidney diseases in children (for trial)Ⅰ. Hormone-sensitive, relapsed/dependent nephrotic syndrome diagnostic and evidence-based guidelines; Ⅲ.Diagnostic criteria for the diagnostic and evidence-based guidelines for hormone-resistant nephrotic syndrome, which means children who are diagnosed with primary nephrotic syndrome should be included;
2. Age from 1 to18;
3. ALT and AST levels do not exceed twice the upper limit of the normal range;;
4. Provision of written informed consent by legal guardians.

Exclusion Criteria:

1. a variety of secondary nephrotic syndromes are caused by infectious diseases such as lupus nephritis, hepatitis b associated nephritis, purpura nephritis, and EB virus, cytomegalovirus (CMV), etc;
2. with combined diseases of cardiovascular, liver, hematopoietic system, mental disorders and other serious diseases;
3. History of diabetes or examinations showed elevated blood glucose levels;
4. Participation in other ongoing clinical trials or during their observation period within the last three months prior to visit 1;
5. Previous/concomitant treatment with any other immunomodulators within the last three months prior to visit 1 ;
6. Patients who are unlikely to adhere to the protocol.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children are diagnosed with primary nephrotic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 1507 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Duration of positive urine protein test changing to the negative result | 48 weeks after treatment
  Duration of positive urine protein test changing to the negative result was measured from day 1 until the time of positive urine protein test changing to negative, assessed up to 48 weeks.
The ratio of positive to negative urine protein | 48 Weeks after treatment
  The proportion of negative urine protein subjects to the total number of subjects, measured from day 1 until the time of positive urine protein test changing to negative, assessed up to 48 weeks.
The decrease of 24-hour urine protein level | 48 Weeks after treatment
  Compared 24-hour urine protein level between baseline and follow-up timepoint, measured from day 1 until time of positive urine protein test changing to negative, assessed up to 48 weeks.

SECONDARY OUTCOMES:
Recovery of blood albumin levels | 48 Weeks after treatment
  Compared blood albumin levels between baseline and follow-up timepoint, assessed up to 48 weeks.
Recurrence rate of PNS | 48 Weeks after treatment
  The proportion of recurrent subjects to the total number of subjects.
Rates of infectious complications of PNS | 48 Weeks after treatment
  The proportion of complicated infectious subjects to the total number of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Chaoying Chen, Professor, Principal Investigator — Children's Hospital of The Capital Institute of Pediatrics
Locations (17):
- China (17):
  - Children's Hospital Capital Institute Of Pediatrics, Beijing, Beijing Municipality
  - Harbin Children's Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Weihui, Henan
  - Henan Children's Hospital, Zhengzhou, Henan
  - Benq Medical Center, Nanjing, Jiangsu
  - Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi Children's Hospital, Wuxi, Jiangsu
  - Xuzhou Children's Hospital, Xuzhou, Jiangsu
  - Jiangxi Provincal Children's Hospital, Nanchang, Jiangxi
  - The first Bethune Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Children's Hospital of Shanxi, Taiyuan, Shanxi
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Urumqi first people's Hospital, Ürümqi, Xinjiang
  - Children's Hospital of Chongqing Medical University, Chongqing
  - Tianjin Children's Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No